CLINICAL TRIAL: NCT05739058
Title: Violet-Blue Light Inactivation of Bacteria in Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Hvidovre University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Frederik Plum, MD, Ph.D Fellow at University of Copenhagen, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: Violet-Blue-Light-Inactivation
Record Dates: First submitted 2023-01-12; First posted 2023-02-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Phototherapy Complication; Photobiology; Light Treatment; Complications; Wound Infection; Wound Heal
Keywords: Violet Blue Light; Blue Light; Safety
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Intervention Model Description: This four-week prospective clinical investigation will assess the safety and feasibility of a medical device emitting LED violet-blue light. Violet-blue light treatment is tested on a total of twenty-two patients with chronic wounds, divided into three groups, each group only receiving one dosage. Three dosages (low, medium and high) of violet-blue light treatment is tested. ID 1-7 are assigned to the low group, ID 8-15 are assigned to medium group and ID 16-22 are assigned to the high dosage group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Exposure to Violet-Blue Light (Experimental): ID 1-7 are assigned to the low dosage group
  Interventions: Device: Violet-Blue Light Treatment / FlashHeal Device
- Medium Exposure to Violet-Blue Light (Experimental): ID 8-15 are assigned to the medium dosage group
  Interventions: Device: Violet-Blue Light Treatment / FlashHeal Device
- High Exposure to Violet-Blue Light (Experimental): ID 16-22 are assigned to the high dosage group
  Interventions: Device: Violet-Blue Light Treatment / FlashHeal Device

INTERVENTIONS:
Device: Violet-Blue Light Treatment / FlashHeal Device — FlashHeal illuminates an area of 10 cm in diameter, located at 6-7 cm distance of the wound.
  Wounds larger than 10 cm in diameter, will receive enough treatments to cover the wound bed.
  To obtain full coverage the circular treatment area is relocated to cover the remaining wound field.
  The wavelength is 405 nm, Full Width Half Maximum at (FWHM) 400-415 nm. Device irradiances are adjusted to the total fluences required for the Low, Medium and High group, the treatment will last 15 minutes at all dosages. Light is emitted with 1000 Hz.

SUMMARY:
This four-week prospective clinical investigation will assess the safety and feasibility of a medical device without CE-marking. The medical device is a light-emitting-diode (LED) and is manufactured by VulCur MedTech Aps. Violet-blue light treatment is tested on a total of twenty-two patients with chronic wounds, divided into three groups, each group only receiving one dosage. Three dosages (low, medium and high) of violet-blue light treatment is tested. ID 1-7 are assigned to the low group, ID 8-15 are assigned to medium group and ID 16-22 are assigned to the high dosage group.

DETAILED DESCRIPTION:
This is as prospective safety and feasibility clinical trial investigating violet-blue light treatment on chronic wounds. This clinical trial runs from Q3 2022 - Q2 2023. Twenty-two patients with chronic wounds will be included (n = 22) for a study-period of four weeks. Week 1 includes one baseline visit. Through Week 2,3 and 4 treatment is given six times with a span of 24-72 hours between every treatment visit. Week 4 includes one follow up-visit. Patients entering the study are assigned to three light dosage groups (low, medium and high) according to their study ID. ID 1-7 are assigned to the low group, ID 8-15 are assigned to medium group and ID 16-22 are assigned to the high dosage group. Between each dosage of light, there will be an evaluation of primary and secondary endpoints by the sponsor and the principal investigator. Light dosage is only escalated should this evaluation be deemed safe. To determine treatment safety skin reactions are assessed after treatment at: 0 minutes, 30 minutes, 24 hours, 48 hours, 5th treatment visit and at follow-up. Adverse Events and Adverse Device Events are evaluated at every visit for every dosage, feasibility is evaluated at follow-up for both patient and investigator. This investigation complies with the Good Clinical Practice concerning medical devices and follows the ISO standard DS/EN 14 155 and the Declaration of Helsinki

ELIGIBILITY:
Inclusion Criteria:

* Men, women and non-binaries fulfilling all inclusion criteria
* Age >18 - Patients with a chronic wound defined > 6 weeks
* Wound Area > 1 cm and < 25 cm
* Patient can understand Danish
* Patient can comply with protocol
* Patient is fully informed about the study and has given informed consent

Exclusion Criteria:

* Clinical infection in the wound requiring systemic or local antibiotics
* Current intake of antibiotics or locally applied (within 7 days before baseline)
* Known or suspected cancer in the wound
* Previous Photodermatitis and/or Photosensitivity
* Previous Porphyria and/or hypersensitivity to porphyrins
* Known congenital or acquired immunodeficiency
* Newly adjusted or newly started systemic immunomodulate treatment >4 weeks
* Treatment with haemodialysis
* Dementia - Participating in other clinical wound healing studies in the last 30 days
* Judgement by the investigator that the patient is not suited for study participation
* Pregnant or breastfeeding women. (All fertile women who is not on safe contraception will need a negative pregnancy test performed at baseline. Safe contraception includes cobber and hormone Intra Uterine Device and Hormone anticonception drugs. Sterility is defined as have had surgical sterilisation and being postmenopausal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are included based on self-representation of gender identity, including non-binary self-representation.
Enrollment: 22 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Overall Common Terminology Criteria for Adverse Events, version 5.0, Nov 27, 2017 (CTCAE) | 4 weeks
  Safety is measured as the absence of Adverse Events (AE) skin reactions. Adverse event skin reactions are assessed with the Common Terminology Criteria for Adverse Events U.S Department of Health and Human Services version 5.0, Nov 27, 2017 (CTCAE) adjusted to the skin. The violet-blue light treatment will be considered safe when less than 30 % have an overall CTCAE score larger than Grade 2 CTCAE. The overall CTCAE score for each patient is based on the one CTCAE score with the most severe grading.

SECONDARY OUTCOMES:
Baseline Clinical Wound Assessment | Baseline, 1 week
  Evaluates wound symptoms (Exudate, necrosis, maceration, granulation, Oedema,) and skin symptoms (eczema, Erythema, Hyperpigmentation, Hypopogmentation, epthilializing) at a 4 step scale from none to mild, moderate, severe.
Clinical Wound Assessment | Pre-intervention, up to 3 weeks
  Evaluates wound symptoms (Exudate, necrosis, maceration, granulation, Oedema,) and skin symptoms (eczema, Erythema, Hyperpigmentation, Hypopogmentation, epthilializing) at a 4 step scale from none to mild, moderate, severe.
Follow up Clinical Wound Assessment | Follow Up, up to 4 weeks
  Evaluates wound symptoms (Exudate, necrosis, maceration, granulation, Oedema,) and skin symptoms (eczema, Erythema, Hyperpigmentation, Hypopogmentation, epthilializing) at a 4 step scale from none to mild, moderate, severe.
Numeric Rating Scale (1-10) | Post-intervention, up to 3 weeks
  Pain scale in relation to treatment. Higher scores indicate more pain.
Wong Baker FACES (1-10) | Post-intervention, up to 3 weeks
  Visual Pain scale in relation to treatment. Higher scores indicate more pain.
Investigator Questionnaire | 4 weeks
  Usability of the medical device is tested with the system usability Scale (SUS) testing 10 items on a 5 step scale from Strongly Disagree to Strongly Agree.
Patient Questionnaire | 4 weeks
  Evaluating Participant perceived; pain, time consumption and satisfaction through 20 items.
  Question 1-13 can be answered on a 5 step scale from "to a very high degree" till "not at all", including possibility to answer "dont know" and "not relevant".
  Item 14-20 can be answered with "Yes", "No" and "Dont Know".
Mean time of visit | For every visit, up to 4 weeks
  Total time for the visit will be measured in minutes.
Mean time of Treatment Procedure | Post-intervention, up to 3 weeks
  For every treatment visit, time used for the treatment with the FlashHeal Device is measured.
  Time is measured in minutes.
Baseline Mean Bacterial Load | 1 week
  E-Swabs, Essen Rotary Technique performed at baseline, follow-up and before and after treatment with FlashHeal Device. Bacteria will be cultured for aerobe and anaerobe species.
Pre-intervention Mean Bacterial Load | Pre-intervention, up to 3 weeks
  E-Swabs, Essen Rotary Technique performed at baseline, follow-up and before and after treatment with FlashHeal Device. Bacteria will be cultured for aerobe and anaerobe species.
Post-intervention Mean Bacterial Load | Post-intervention, up to 3 weeks
  E-Swabs, Essen Rotary Technique performed at baseline, follow-up and before and after treatment with FlashHeal Device. Bacteria will be cultured for aerobe and anaerobe species.
Mean Bacterial Load at Follow Up | Follow up, up to 4 weeks
  E-Swabs, Essen Rotary Technique performed at baseline, follow-up and before and after treatment with FlashHeal Device. Bacteria will be cultured for aerobe and anaerobe species.
Baseline Wound Fluid | Baseline, 1 Week
  Swab for wound fluid performed once every week using the Essen Rotary Technique, testing for 6-10 cytokines assessing the inflammatory microenvironment.
Change from Baseline Wound Fluid Composition Week 1 to Week 2 | 2 Weeks
  Swab for wound fluid performed once every week using the Essen Rotary Technique, testing for 6-10 cytokines assessing the inflammatory microenvironment.
Change from Baseline Wound Fluid Composition Week 1 to Week 3 | 3 Weeks
  Swab for wound fluid performed once every week using the Essen Rotary Technique, testing for 6-10 cytokines assessing the inflammatory microenvironment.
Change from Baseline Wound Fluid Composition Week 1 to Week 4 | 4 weeks
  Swab for wound fluid performed once every week using the Essen Rotary Technique, testing for 6-10 cytokines assessing the inflammatory microenvironment.
Baseline Wound Size Week 1 | Baseline, week 1
  Clinical Photography is performed once every week. Hereafter the wound is analysed with the ImageJ software to calculate wound size in cm2.
Change from Baseline Wound Size Week 1 to Week 2 | 2 Weeks
  Clinical Photography is performed once every week. Hereafter the wound is analysed with the ImageJ software to calculate wound size in cm2.
Change from Baseline Wound Size Week 1 to Week 3 | 3 Weeks
  Clinical Photography is performed once every week. Hereafter the wound is analysed with the ImageJ software to calculate wound size in cm2.
Change from Baseline Wound Size Week 1 to Week 4 | Follow Up, 4 weeks
  Clinical Photography is performed once every week. Hereafter the wound is analysed with the ImageJ software to calculate wound size in cm2.
Common Terminology Criteria for Adverse Events, version 5.0, Nov 27, 2017 (CTCAE) | Post-intervention, 2 weeks
  Safety is measured as the absence of Adverse Events (AE) skin reactions. Adverse event skin reactions are assessed with the Common Terminology Criteria for Adverse Events U.S Department of Health and Human Services version 5.0, Nov 27, 2017 (CTCAE). The CTCAE is adjusted to the skin.
Common Terminology Criteria for Adverse Events, version 5.0, Nov 27, 2017 (CTCAE) | 30 minutes Post-intervention, 2 weeks
  Safety is measured as the absence of Adverse Events (AE) skin reactions. Adverse event skin reactions are assessed with the Common Terminology Criteria for Adverse Events U.S Department of Health and Human Services version 5.0, Nov 27, 2017 (CTCAE). The CTCAE is adjusted to the skin.
Common Terminology Criteria for Adverse Events, version 5.0, Nov 27, 2017 (CTCAE) | 24 hours Post-intervention, 2 weeks
  Safety is measured as the absence of Adverse Events (AE) skin reactions. Adverse event skin reactions are assessed with the Common Terminology Criteria for Adverse Events U.S Department of Health and Human Services version 5.0, Nov 27, 2017 (CTCAE). The CTCAE is adjusted to the skin.
Common Terminology Criteria for Adverse Events, version 5.0, Nov 27, 2017 (CTCAE) | 48 hours Post-intervention, 2 weeks
  Safety is measured as the absence of Adverse Events (AE) skin reactions. Adverse event skin reactions are assessed with the Common Terminology Criteria for Adverse Events U.S Department of Health and Human Services version 5.0, Nov 27, 2017 (CTCAE). The CTCAE is adjusted to the skin.
Common Terminology Criteria for Adverse Events, version 5.0, Nov 27, 2017 (CTCAE) | 120 hours Post-intervention, 2 weeks
  Safety is measured as the absence of Adverse Events (AE) skin reactions. Adverse event skin reactions are assessed with the Common Terminology Criteria for Adverse Events U.S Department of Health and Human Services version 5.0, Nov 27, 2017 (CTCAE).
  The CTCAE is adjusted to the skin.
Common Terminology Criteria for Adverse Events, version 5.0, Nov 27, 2017 (CTCAE) | Follow Up, 4 weeks
  Safety is measured as the absence of Adverse Events (AE) skin reactions. Adverse event skin reactions are assessed with the Common Terminology Criteria for Adverse Events U.S Department of Health and Human Services version 5.0, Nov 27, 2017 (CTCAE).
  The CTCAE is adjusted to the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Plum, MD, Principal Investigator — Danish Wound Healing Center, Bispebjerg Hospital
Locations (1):
- Danish Wound Healing Center, Bispebjerg Hospital, Copenhagen, Northwest, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjarnsholt T, Kirketerp-Moller K, Jensen PO, Madsen KG, Phipps R, Krogfelt K, Hoiby N, Givskov M. Why chronic wounds will not heal: a novel hypothesis. Wound Repair Regen. 2008 Jan-Feb;16(1):2-10. doi: 10.1111/j.1524-475X.2007.00283.x. PMID 18211573
- [Background] Malone M, Bjarnsholt T, McBain AJ, James GA, Stoodley P, Leaper D, Tachi M, Schultz G, Swanson T, Wolcott RD. The prevalence of biofilms in chronic wounds: a systematic review and meta-analysis of published data. J Wound Care. 2017 Jan 2;26(1):20-25. doi: 10.12968/jowc.2017.26.1.20. PMID 28103163
- [Background] Enwemeka CS. Antimicrobial blue light: an emerging alternative to antibiotics. Photomed Laser Surg. 2013 Nov;31(11):509-11. doi: 10.1089/pho.2013.9871. Epub 2013 Oct 18. No abstract available. PMID 24138170
- [Background] Leanse LG, Dos Anjos C, Mushtaq S, Dai T. Antimicrobial blue light: A 'Magic Bullet' for the 21st century and beyond? Adv Drug Deliv Rev. 2022 Jan;180:114057. doi: 10.1016/j.addr.2021.114057. Epub 2021 Nov 18. PMID 34800566
- [Background] Tomb RM, White TA, Coia JE, Anderson JG, MacGregor SJ, Maclean M. Review of the Comparative Susceptibility of Microbial Species to Photoinactivation Using 380-480 nm Violet-Blue Light. Photochem Photobiol. 2018 May;94(3):445-458. doi: 10.1111/php.12883. Epub 2018 Mar 31. PMID 29350751
- [Background] Plattfaut I, Demir E, Fuchs PC, Schiefer JL, Sturmer EK, Bruning AKE, Oplander C. Characterization of Blue Light Treatment for Infected Wounds: Antibacterial Efficacy of 420, 455, and 480 nm Light-Emitting Diode Arrays Against Common Skin Pathogens Versus Blue Light-Induced Skin Cell Toxicity. Photobiomodul Photomed Laser Surg. 2021 May;39(5):339-348. doi: 10.1089/photob.2020.4932. PMID 33961502
- [Background] Dai T, Gupta A, Huang YY, Yin R, Murray CK, Vrahas MS, Sherwood ME, Tegos GP, Hamblin MR. Blue light rescues mice from potentially fatal Pseudomonas aeruginosa burn infection: efficacy, safety, and mechanism of action. Antimicrob Agents Chemother. 2013 Mar;57(3):1238-45. doi: 10.1128/AAC.01652-12. Epub 2012 Dec 21. PMID 23262998
- [Background] Wang Y, Wang Y, Wang Y, Murray CK, Hamblin MR, Hooper DC, Dai T. Antimicrobial blue light inactivation of pathogenic microbes: State of the art. Drug Resist Updat. 2017 Nov;33-35:1-22. doi: 10.1016/j.drup.2017.10.002. Epub 2017 Oct 13. PMID 29145971
- [Background] Liebmann J, Born M, Kolb-Bachofen V. Blue-light irradiation regulates proliferation and differentiation in human skin cells. J Invest Dermatol. 2010 Jan;130(1):259-69. doi: 10.1038/jid.2009.194. PMID 19675580